CLINICAL TRIAL: NCT05342077
Title: Virtual Reality-Reward Training for Anhedonia
Acronym: VR-RT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Michelle Craske, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Virtual Reality Training Study
Record Dates: First submitted 2022-03-16; First posted 2022-04-22 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2024-05

CONDITIONS: Positive Affect; Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual Reality-Reward Training (VR-RT) (Experimental): 7 sessions of positive VR immersion and positive memory specificity training exercises designed to savor rewarding features of immersion followed by memory specificity training exercises to savor rewarding features of autobiographical memory.
  Interventions: Behavioral: Virtual Reality-Reward Training (VR-RT)
- Virtual Reality-Memory Training (VR-MT) (Active Comparator): 7 sessions of neutral VR immersion and neutral memory specificity training exercises, designed to train memory of objective non-emotional stimuli followed by memory exercises to neutral autobiographical memories.
  Interventions: Behavioral: Virtual Reality-Memory Training (VR-MT)

INTERVENTIONS:
Behavioral: Virtual Reality-Reward Training (VR-RT) — Participants will complete verbal recounting (present-tense, field perspective, positive details) and guided imaginal recounting of positive details for rewarding VR experiences and positive autobiographical memories.
  Arms: Virtual Reality-Reward Training (VR-RT)
Behavioral: Virtual Reality-Memory Training (VR-MT) — Participants will complete verbal recounting (past-tense, observer perspective, objective details) and guided imaginal recounting of neutral details for neutral VR experiences and neutral autobiographical memories.
  Arms: Virtual Reality-Memory Training (VR-MT)

SUMMARY:
The purpose of this study is to compare the effects of Virtual Reality-Reward Training (VR-RT) with an active control condition, Virtual Reality-Memory Training (VR-MT), on positive affect and other clinical symptoms.

VR-Reward Training is a novel intervention aimed at enhancing savoring of positive experiences among individuals with depression and low positive affect through guided imaginal recounting following immersion in positive VR experiences.

Target enrollment is 80 male and female participants with low positive affect, depression, and impaired functioning, who are at least 18 years old, who will be randomly assigned to 7 weeks of either Virtual Reality-Reward Training (VR-RT) or Virtual Reality-Memory Training (VR-MT). Participants will complete in-person VR sessions, laboratory assessments, self-report questionnaires as part of the study.

The total length of participation is around 3 months.

DETAILED DESCRIPTION:
Anhedonia, or loss of interest and pleasure in usual activities, has been relatively resistant to pharmacological and psychological treatments in the context of anxiety and depression. Newer treatments that focus upon positivity or reward sensitivity have shown promising results.

The purpose of the current randomized controlled trial is to compare the effects of Virtual Reality-Reward Training (VR-RT) with an active control condition, Virtual Reality-Memory Training (VR-MT), on positive affect and other clinical symptoms. Virtual Reality-Reward Training is designed to augment reward sensitivity in individuals with depression and low positive affect. Targets include behavioral, cognitive, and self-report indices of reward anticipation and initial response to reward. Specificity of target engagement is assessed by comparison with Virtual Reality-Memory Training, designed to improve memory.

Targets and clinical outcomes are assessed at baseline (Week 1) and either weekly or at mid-treatment (Week 3), post-treatment (Week 7), and follow-up (Week 12). Statistical models evaluate whether change in outcomes and change in target measures are greater as a result of Virtual Reality-Reward Training compared to Virtual-Reality-Memory Training and whether changes in target measures correlate with changes in outcome measures.

Target enrollment is 80 male and female participants with low positive affect, depression, and impaired functioning, who are at least 18 years old, who will be randomized to Virtual Reality-Reward Training or Virtual-Reality Memory Training, each comprising 7 individual virtual reality training sessions over the course of 7 weeks.

Participants will complete laboratory tests and self-report questionnaires as part of the study. Total length of participation is around 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old
2. Fluent in written and spoken English
3. Meet all of the following dimensional score cutoffs:

   1. Score on the DASS-21 depression subscale must be ≥ 11
   2. Score on the PANAS-P of 24 or lower
   3. Score on the SDS of ≥ 6
4. Willingness to refrain from initiating other psychosocial treatments throughout the duration of the study

Exclusion Criteria:

1. Lifetime history of bipolar disorder, psychosis, mental retardation, or organic brain damage
2. Substance use disorder in the past 6 months
3. Current use of psychotropic medications
4. Currently pregnant or planning to become pregnant
5. Self-reported frequent motion sickness
6. Self-reported seizures within the last year and/or a diagnosis of epilepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2025-03-14 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
Depression, Anxiety, and Stress Scales (DASS-21) | Change from baseline to follow-up (Week 12)
  Reported symptoms of depression (score range: 0-21), anxiety (score range: 0-21), and stress (score range: 0-21), higher scores indicate higher severity and frequency.
The Positive Affect and Negative Affect Schedule-Expanded Form (PANAS X) (General Dimensions Scales) | Change from baseline to follow-up (Week 12)
  Change in reported positive affect (general dimensions scale positive affect) and negative affect (general dimension scale negative affect) (score range for each scale: 10-50, higher scores represent higher levels of positive affect or negative affect).
MASQ-AD 14 Item | Change from baseline to follow-up (Week 12)
  Change in reported anhedonia (score range: 14-70), with higher scores indicating greater anhedonic symptom severity

SECONDARY OUTCOMES:
Behavioral Activation Scale (BAS) | Change from baseline to follow-up (Week 12)
  Change in reported reward sensitivity (score range: 23-92), with higher scores indicating higher reward sensitivity
Work and Social Functioning Scale (WSAS) | Change from baseline to follow-up (Week 12)
  Change in impairment in the following life domains: work (score range: 0-8), home management (score range: 0-8), social leisure (score range: 0-8), private leisure (score range: 0-8) and personal or family relationships (score range: 0-8).
Positive and Negative Affective Schedule (PANAS) | Change from baseline to follow-up (Week 12)
  Change in reported positive affect and negative affect (score range for each scale: 10-50, higher scores indicate higher levels of positive affect or negative affect)
Temporal Experience of Pleasure Scale (TEPS) | Change from baseline to follow-up (Week 12)
  Change in reported anticipatory pleasure (score range: 10-60) and consummatory pleasure (score range: 8-48). Higher scores indicate higher reward responsiveness.
Effort Reward Trade-off Task | Change from baseline to follow-up (Week 12)
  Change in behavioral effort for reward (button presses for points) and experience of reward (happiness ratings). The Effort Reward Trade-off Task is a novel online behavioral task.
Positive Valence Systems Scale (PVSS-21) | Change from baseline to follow-up (Week 12)
  Change in reward anticipation, motivation, and consumption for rewards such as rewards such as food, physical touch, positive feedback, social interactions, hobbies and goals (score range: 21-105). Higher scores (e.g. 105) indicate higher reward responsiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle G Craske, Ph.D, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No